CLINICAL TRIAL: NCT00424970
Title: Hypoventilation and High Altitude Chronic Polycythemia: Acetazolamide as a Possible Treatment
Brief Title: Treatment of High Altitude Polycythemia by Acetazolamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association pour la Recherche en Physiologie de l'Environnement (Other)
Collaborators: University of Paris 13 (Other); Universidad Peruana Cayetano Heredia (Other); Legs Poix (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APCA06; Legs Poix 999
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: High Altitude Polycythemia
Keywords: high altitude; hypoxia; pulmonary hypertension; polycythemia; hypoventilation
MeSH Terms: conditions — Altitude Sickness; Hypoxia; Hypertension, Pulmonary; Polycythemia; Hypoventilation | interventions — Acetazolamide

ARMS (1):
- acetazolamide (Placebo Comparator): acetazolamide 250mg /day oral administration, for 6 months
  Interventions: Drug: acetazolamide

INTERVENTIONS:
Drug: acetazolamide

SUMMARY:
The prevalence of High Altitude Polycythemia (or Chronic Mountain Sickness) is between 8 and 15% in the high altitude regions of South America. There is no pharmacological treatment available. After a first preliminary study in 2003 demonstrating the beneficial effects of acetazolamide in reducing hematocrit in these patients, after 3 weeks of treatment, we want to confirm this effect and implement a treatment protocol of 3 month-duration.

DETAILED DESCRIPTION:
Chronic mountain sickness (CMS) is characterized by an excessive number of red cells in the blood of persons living permanently above the altitude of 2,500m. The symptoms of this very incapacitating disease are : headaches, chronic asthenia, digestive troubles, sleep disturbances. The hemoglobin concentration is higher than 21 g/dl of blood. In addition, patients show a pulmonary hypertension of variable degree, as well as a systemic hypertension.

This disease affects essentially males, but women are also concerned after menopause. The evolution of the disease is always very dramatic, towards a cardiac failure and cerebral vascular stroke. The prevalence is between 8% and 15% on the Andean Altiplano . No pharmacological treatment is available.

A preliminary study was performed (Richalet et al. AJRCCM, 2005) that demonstrated the efficiency of acetazolamide (a carbonic anhydrase inhibitor) in reducing the hematocrit and the erythropoetin concentration,and increasing nocturnal oxygen saturation in patients suffering from CMS, after 3 weeks of treatment.

We plan to perform a double-blinded placebo-controlled study to evaluate the efficiency of a 3-month treatment with daily 250 mg acetazolamide to reduce the hematocrit and hemoglobin concentrations and ameliorate the clinical symptoms of 55 patients suffering from CMS and living at high altitude (Cerro de Pasco, Peru).

ELIGIBILITY:
Inclusion Criteria:

* patients with Chronic mountain sickness and Hb > 21g/dl

Exclusion Criteria:

* patients smokers
* patients with respiratory or cardiovascular or renal disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2007-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration | monthly
Hematocrit | monthly

SECONDARY OUTCOMES:
Systolic pulmonary arterial pressure | before and after 3 months of treatment
Pulmonary vascular resistance | before and after 3 months of treatment
Arterial oxygen saturation at rest | monthly
Clinical score of Chronic Mountain Sickness | monthly
Quality of lofe score | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Richalet, MD, PHD, Principal Investigator — ARPE, University Paris 13; Fabiola Leon-Velarde, PHD, Study Director — University Cayetano Heredia, Lima, Peru
Locations (1):
- University Cayetano Heredia, Lima, Peru

REFERENCES:
- [Background] Richalet JP, Rivera M, Bouchet P, Chirinos E, Onnen I, Petitjean O, Bienvenu A, Lasne F, Moutereau S, Leon-Velarde F. Acetazolamide: a treatment for chronic mountain sickness. Am J Respir Crit Care Med. 2005 Dec 1;172(11):1427-33. doi: 10.1164/rccm.200505-807OC. Epub 2005 Aug 26. PMID 16126936
- [Derived] Maignan M, Rivera-Ch M, Privat C, Leon-Velarde F, Richalet JP, Pham I. Pulmonary pressure and cardiac function in chronic mountain sickness patients. Chest. 2009 Feb;135(2):499-504. doi: 10.1378/chest.08-1094. Epub 2008 Aug 21. PMID 18719057
- [Derived] Richalet JP, Rivera-Ch M, Maignan M, Privat C, Pham I, Macarlupu JL, Petitjean O, Leon-Velarde F. Acetazolamide for Monge's disease: efficiency and tolerance of 6-month treatment. Am J Respir Crit Care Med. 2008 Jun 15;177(12):1370-6. doi: 10.1164/rccm.200802-196OC. Epub 2008 Apr 3. PMID 18388356